CLINICAL TRIAL: NCT04388072
Title: An Diagnostic Cohort on Applicability and Accuracy of AQP4-Immunoglobulin G Detection Kit in the Diagnosis of Neuromyelitis Optica Spectrum Disorders
Brief Title: An Diagnostic Cohort on AQP4-Immunoglobulin G Detection Kit
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Collaborators: MyBiotech Co. Ltd, China (Unknown); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ning Wang, MD., PhD., Director, First Affiliated Hospital of Fujian Medical University
Other Study IDs: LS2019-004-02
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnostic cohort study could will be use to verify the clinical performance of the AQP4 -immunoglobulin G detection kit and whether it has a good correlation with the clinical diagnosis results. The applicability and accuracy of the kit in clinical diagnosis will be verified according to the measured data.

ELIGIBILITY:
Inclusion Criteria:

1. The patients who were diagnosed with NMOSD , and the cell-based assay was used to determine the AQP4-IgG-seropositive patients;
2. AQP4-IgG is negative in health people with age and sex matching and determined by cell-based assay;
3. Female or male, age 14-80;
4. Patients or authorized family members volunteered to participate in this study and signed informed consent.

Exclusion Criteria:

1. Patients with coagulation disorders;
2. Infection-related encephalitis;
3. Immune-related encephalitis;
4. A patient with severe mental illness who cannot cooperate clinically;
5. A patient with severe jaundice.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with NMOSD who are diagnosied in the First Affiliated Hospital of Fujian Medical Universtiy by two neurolgists
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
results of AQP4 -immunoglobulin G detection kit | through study completion, an average of 6 months
  The Serum test results of participants using AQP4 -immunoglobulin G detection kit

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Neurology,First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Third Affiliated Hospital of Sun Yat-sen University, Guangzhou